CLINICAL TRIAL: NCT07110350
Title: Clinical Characteristics and Outcomes of Non-Indicated Staged Laparotomies in Abdominal Trauma Patients: A Single-Center Retrospective Study
Brief Title: Clinical Outcomes of Non-Indicated Staged Laparotomies in Abdominal Trauma
Status: Not yet recruiting | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: FEMH_Treauma_114107-E
Record Dates: First submitted 2025-07-01; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Abdominal Trauma; Damage Control Surgery; Laparotomy
MeSH Terms: conditions — Abdominal Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- single vs. staged operation: Patients will be categorized based on the number of operations (single vs. staged), and further stratified by whether the initial operation met the criteria for a staged approach.
  Interventions: Procedure: Laparotomy refers to a definitive single-stage exploratory abdominal surgery. Damage Control Surgery refers to a staged surgical approach including initial abbreviated laparotomy followed by planned.

INTERVENTIONS:
Procedure: Laparotomy refers to a definitive single-stage exploratory abdominal surgery. Damage Control Surgery refers to a staged surgical approach including initial abbreviated laparotomy followed by planned. — This intervention involves exploratory laparotomy performed for abdominal trauma at a single tertiary care trauma center in Taiwan between 2013 and 2024. Patients are stratified based on whether they received a single definitive laparotomy or staged damage control surgery. Staged surgery is defined as an abbreviated initial laparotomy followed by planned reoperation(s), regardless of whether physiological indications were strictly met. This study specifically investigates the discrepancy between guideline-based indications and actual surgical practice.

SUMMARY:
The goal of this observational study is to understand how often staged operations are performed in abdominal trauma patients without meeting standard clinical criteria, and to explore related clinical characteristics and outcomes. The main questions it aims to answer are:

How frequently are staged operations performed when not clinically indicated?

What are the clinical features and outcomes of patients who undergo non-indicated staged operations?

What are the risk factors for delayed reoperation among patients who initially received a single operation?

Researchers will review medical records of patients who underwent exploratory laparotomy for abdominal trauma at Far Eastern Memorial Hospital between January 1, 2013, and December 31, 2024. Participants will be grouped based on whether they had a single or staged operation, and whether their initial operation met established criteria for a staged approach. Clinical characteristics and outcomes will be compared across groups.

DETAILED DESCRIPTION:
Background:

Staged operation, a key component of damage control surgery, is typically indicated for trauma patients with physiological instability, including hypotension, hypothermia, metabolic acidosis, or coagulopathy. However, deviations from these criteria are frequently observed in clinical practice, raising concerns about discrepancies between guidelines and surgical decisions, and the potential for overuse.

Objective:

This study aims to investigate the disparity between clinical indications and actual use of staged operations in patients with abdominal trauma, and to explore associated clinical characteristics and possible prognostic implications.

Methods:

A retrospective review will be conducted on patients who underwent exploratory laparotomy for abdominal trauma at Far Eastern Memorial Hospital between January 1, 2013, and December 31, 2024. Patients will be categorized based on the number of operations (single vs. staged), and further stratified by whether the initial operation met the criteria for a staged approach. Among those not meeting the criteria, clinical features and outcomes will be compared. Additionally, risk factors for delayed reoperation in initially single-operation patients will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* This study included patients with abdominal trauma who were admitted to Far Eastern Memorial Hospital and received exploratory laparotomy between January 1, 2013, and December 31, 2024.

Exclusion Criteria:

* Patients who experienced cardiac arrest prior to hospital arrival (OHCA) or in-hospital cardiac arrest (IHCA).
* Patients with an Abbreviated Injury Scale (AIS) score ≥ 4 in any body region other than the abdomen.
* Patients who died within 24 hours after the most recent surgical procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes patients with abdominal trauma who were admitted to Far Eastern Memorial Hospital between January 1, 2013, and December 31, 2024, and underwent exploratory laparotomy. Patients under 18 years of age, those with pre-hospital or in-hospital cardiac arrest, those with an Abbreviated Injury Scale (AIS) score ≥ 4 in non-abdominal regions, and those who died within 24 hours after the latest surgery were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
death | From enrollment to the end of treatment at 6 months
  The primary outcome is defined as all-cause mortality occurring no earlier than 24 hours after the most recent surgical intervention.

SECONDARY OUTCOMES:
Complications | through study completion, an average of 1 year
  Secondary outcomes included postoperative complications such as ileus, infection, poor wound healing, and incisional hernia.

CONTACTS AND LOCATIONS:
Overall Officials: Chien Wu, MD, Principal Investigator — Department of Surgery, Far Eastern Memorial Hospital
Locations (1):
- Far Estern Memorial Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-08-03): https://cdn.clinicaltrials.gov/large-docs/50/NCT07110350/Prot_SAP_000.pdf